CLINICAL TRIAL: NCT05593757
Title: Quinidine Versus Verapamil in Short-coupled Idiopathic Ventricular Fibrillation: an Open-label, Randomized Crossover Pilot Trial
Brief Title: Quinidine Versus Verapamil in Short-coupled Idiopathic Ventricular Fibrillation
Acronym: QUEEN-IVF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Christian van der Werf, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022.0479
Record Dates: First submitted 2022-10-10; First posted 2022-10-25 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Short-coupled Idiopathic Ventricular Fibrillation
MeSH Terms: interventions — Quinidine; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quinidine in period A, verapamil in period B (Experimental): For this arm, patients will be treated with quinidine 200 mg thrice daily during period A. During period B, patients will be treated with verapamil 320-480mg daily during period B. The duration of the periods is different for each patient and depends on the time of inclusion.
  Interventions: Drug: Quinidine; Drug: Verapamil
- Verapamil in period A, quinidine in period B (Experimental): For this arm, patients will be treated with verapamil 320-480mg daily during period A. During period B, patients will be treated with quinidine 200 mg thrice daily during period A. The duration of the periods is different for each patient and depends on the time of inclusion.
  Interventions: Drug: Quinidine; Drug: Verapamil

INTERVENTIONS:
Drug: Quinidine — Oral quinidine
Drug: Verapamil — Oral verapamil

SUMMARY:
Short-coupled idiopathic ventricular fibrillation (IVF) is a rare subtype of idiopathic ventricular fibrillation that is characterized by ventricular fibrillation (VF) or polymorphic ventricular tachycardia (PVT) initiated by a short-coupled premature ventricular contraction (PVC). Although patients are protected from sudden cardiac death by an implantable cardioverter-defibrillator (ICD), additional antiarrhythmic drug therapy is indispensable as recurrent ICD shocks are not uncommon and can negatively affect quality of life. Verapamil and quinidine have been suggested as effective antiarrhythmic drugs, but at present it is unknown whether these drugs reduce the incidence of arrhythmic events. This pilot study will provide insight into the advisability and feasibility of a randomized controlled trial (RCT) and provide data needed to determine the most appropriate design and the sample size.

ELIGIBILITY:
Inclusion Criteria:

1. At least one of the following 3 principal diagnostic criteria for short-coupled IVF:

   A. Diagnosis of short-coupled IVF, based on any documentation (i.e., ECG, Holter monitor, device electrogram (EGM), or telemetry) of PVT of ≥3 consecutive beats or VF initiated by a PVC with a coupling interval <350 ms B. Isolated PVCs with a coupling interval <350 ms during the index admission after SCA based on a shockable rhythm or (presumed) arrhythmogenic syncope C. DPP6 haplotype carrier
2. Functioning transvenous or subcutaneous ICD in place
3. Sudden cardiac arrest, (near)syncope, appropriate ICD shock or nonsustained PVT documented by the ICD at least once in the past 2 years
4. Genetic testing has been initiated. Results are not required to be known at the time of inclusion. In subjects who are family members of DPP6 carrying index patients, genes other than DPP6 are not required to be tested
5. Willing to undergo two assigned treatment periods with verapamil and quinidine
6. Age ≥ 18 years

Exclusion Criteria:

* Pregnancy or lactation
* Current treatment with class 1 antiarrhythmic medication (other than quinidine), class 3 antiarrhythmic medication, or digoxin, unless this medication is discontinued; patients who are currently treated with amiodarone will not be included due to the long elimination half-life of amiodarone, unless amiodarone was only administered intravenously for a short period of time
* Patients with a history of therapy refractory ventricular arrhythmia on an adequate dose of verapamil or quinidine, as determined by the treating cardiologist.
* Contra-indication to quinidine or verapamil (see section 7.6)
* Significant structural heart disease (left ventricular ejection fraction <50%, suspicion or definitive diagnosis of cardiomyopathy, moderate/severe pulmonary, mitral, or aortic valve stenosis or regurgitation)
* Suspicion or definitive diagnosis of another (heritable) arrhythmia syndrome, e.g.

Brugada syndrome, early repolarization syndrome or catecholaminergic polymorphic ventricular tachycardia

* Presence of a short (<350 ms) or prolonged (>480 ms) heart-rate corrected QT interval on the resting ECG at baseline
* Presence of a pathogenic or likely-pathogenic ryanodine receptor 2 (RYR2) mutation
* Presence of ischemia-induced short-coupled ventricular arrhythmia in patient with documented coronary spasm
* Presence of pause-dependent torsade de pointes [preceding R-R interval prior to the trigger PVC >1500 ms in individuals without pacemaker/ICD or >1300 ms in individuals with pacemaker/ICD] following a stable baseline rhythm. Initiation of ventricular arrhythmia by short-long-short cycles (R-R cycles <1300 ms) with a short-coupled trigger PVC is allowed
* Significant coronary artery disease (≥50% narrowing of the diameter of the lumen of the left main coronary artery or ≥70% narrowing of the diameter of the lumen of the left anterior descending coronary artery, left circumflex artery or right coronary artery)
* Reversible metabolic or pharmacological/toxicological conditions that may cause electrophysiological findings similar to short-coupled IVF
* Patients who are considered electrically unstable, at physician's discretion, due to active electrical storm or very frequent nonsustained episodes of short-coupled IVF requiring intravenous or invasive therapy
* Successful radiofrequency ablation of the PVC initiating short-coupled IVF and absence of documented (non)sustained episodes of short-coupled PVT/VF afterwards. The patient will, however, be eligible to participate in the study if ≥ 1 episode of short-coupled PVT/VF is documented after the ablation procedure
* Intention to perform radiofrequency ablation of the PVC initiating short-coupled IVF during the course of the study
* Serious known comorbid disease with a life expectancy of less than two years
* Ongoing medical condition that is deemed by the principal investigator to interfere with the conduct or assessments of the study or safety of the subjects
* Circumstances that prevent follow-up
* Inability to take orally administered tablets
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Sustained ventricular arrhythmia | 3 years
  Sustained ventricular arrhythmia, assessed using the severity scoring system. A subject will be scored in each treatment period according to the scoring system by the Endpoint Classification Committee. The highest applicable score will be used.
  Ventricular arrhythmia scoring system:
  0= No arrhythmic events
  1. A single arrhythmic event
  2. Electrical storm (≥3 episodes of sustained PVT/VF within 24 hours)
  3. ≥2, but <5 arrhythmic events
  4. ≥5 arrhythmic events

SECONDARY OUTCOMES:
Time to first arrhythmic event | 3 years
  The time between the first day in each period and the first arrhythmic event in that period
Incidence of quinidine-induced torsade de pointes | 3 years
Incidence of sustained monomorphic ventricular tachycardia | 3 years
Number of inappropriate ICD shocks | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian van der Werf, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands